CLINICAL TRIAL: NCT00527501
Title: IOP Lowering Efficacy of Travoprost/Brinzolamide Fixed Combination Ophthalmic Suspension in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-07-07
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2008-02

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: Open-angle glaucoma; ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost; brinzolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Travoprost/brinzolamide

SUMMARY:
The purpose of this study is to compare the safety and IOP-lowering efficacy of a fixed combination of Travoprost/Brinzolamide Ophthalmuc Suspension dosed BID and QD, to TRAVATAN dosed QD and a Vehicle dosed BID in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older of either sex and any race with diagnosed open-angle glaucoma or confirmed ocular hypertension

Exclusion Criteria:

* Age (Under 18)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Mean IOP | Time

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Landry, Study Director — Alcon Research
Locations (1):
- Artesia, Artesia, California, United States